CLINICAL TRIAL: NCT00878254
Title: Phase II Study of Rituximab in Combination With Methotrexate, Doxorubicin, Cyclophosphamide, Leucovorin, Vincristine, Ifosfamide, Etoposide, Cytarabine and Mesna (R-MACLO/IVAM) in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Previously Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Izidore Lossos, MD, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080803; SCCC-2008043 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Mantle-Cell Lymphoma
Keywords: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Mesna; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- R-MACLO/IVAM Group (Experimental): Participants in this group will receive four 21-day cycles of combination R-MACLO/IVAM induction therapy, followed by Rituximab maintenance therapy as follows:
  Induction Therapy:
  * Cycles 1 and 3: Rituximab, Doxorubicin, Vincristine, Cyclophosphamide, Methotrexate, Leucovorin and Granulocyte-colony stimulating factor (G-CSF)
  * Cycles 2 and 4: Rituximab, Cytarabine, Ifosfamide, Mesna, Etoposide, and G-CSF.
  Maintenance Therapy: Rituximab: For study participants in complete remission. Every 6 months for up to 3 years.
  Total participation duration is about 4 years. Participants will be followed for survival.
  Interventions: Biological: G-CSF; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Doxorubicin; Drug: Etoposide; Drug: Ifosfamide; Drug: Leucovorin; Drug: Mesna; Drug: Methotrexate; Drug: Vincristine

INTERVENTIONS:
Biological: G-CSF — Granulocyte-colony stimulating factor (G-CSF) 480 mcg subcutaneously starting on Day 13 of Cycles 1 and 3; and Day 7 of Cycles 2 and 4.
  Other Names: Filgrastim; Neupogen
Drug: Rituximab — Rituximab 375 mg/m^2 intravenously (IV) on Day 1 for 4 Cycles during induction therapy. Participants achieving complete remission will then receive Rituximab maintenance therapy every 6 months for up to three years.
  Other Names: Rituxan
Drug: Cyclophosphamide — Cyclophosphamide 800 mg/m^2 IV on Day 1 and 200 mg/m^2 IV on Days 2 through 5 of Cycles 1 and 3.
  Other Names: Cytoxan
Drug: Cytarabine — Cytarabine (AraC) 2 grams/m^2 IV on Days 1 and 2 of Cycles 2 and 4.
  Other Names: AraC
Drug: Doxorubicin — Doxorubicin 45 mg/m^2 IV bolus on Day 1 of Cycles 1 and 3.
  Other Names: Adriamycin
Drug: Etoposide — Etoposide (VP16) 60 mg/m^2 IV on Days 1 through 5 of Cycles 2 and 4.
  Other Names: VP16
Drug: Ifosfamide — Ifosfamide 1.5 grams/m^2 IV on Days 1 through 5 of Cycles 2 and 4.
  Other Names: Ifex
Drug: Leucovorin — Leucovorin 100 mg/m^2 IV beginning 36 (+/-4) hours after start of Methotrexate infusion, and then 10 mg/m^2 at 6 hour (+/- 30 min) intervals until Methotrexate level is < 0.1 µmol/L during Cycles 1 and 3.
  Other Names: Folinic acid
Drug: Mesna — Mesna 360 mg/m^2 IV on Days 1 through 5 of Cycles 2 and 4.
  Other Names: Mesnex
Drug: Methotrexate — Methotrexate (MTX) 1,200 mg/m^2 in 250 mL with Dextrose 5% in water (D5W) IV over 1 hour, followed by Methotrexate 3,000 mg/m^2 in 1,000 mL D5W by continuous infusion over 23 (+/-2) hours on Day 10 of Cycles 1 and 3.
  Other Names: MTX
Drug: Vincristine — Vincristine 1.5 mg/m^2 IV push (maximum of 2 mg) on Days 1 and 8 of Cycles 1 and 3.
  Other Names: Oncovin

SUMMARY:
The investigator(s) hypothesize that Rituximab together with combination chemotherapy, followed by Rituximab maintenance therapy, will provide better disease control with improved response rates and overall survival in patients with previously untreated Mantle Cell Lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated, histologically confirmed mantle cell lymphoma,
2. Measurable or evaluable disease (at least one site with >1.5 cm in diameter
3. All stages are eligible
4. Age > 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
6. Adequate hepatic function:

   * Bilirubin < 3 mg/dL
   * Transaminases (serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamate-pyruvate transaminase (SGPT)) < than 2.5 times the upper limit of normal for the institution, unless due to lymphomatous involvement
7. Serum creatinine< 1.5 mg/dl
8. Ability to give informed consent
9. Women of childbearing potential must have a negative pregnancy test within 72 hours of entering into the study. Males and females must agree to use adequate birth control if conception is possible during the study. Women must avoid pregnancy and men avoid fathering children while in the study.
10. Life expectancy greater than 6 months.

Exclusion Criteria:

1. Previous chemotherapy, immunotherapy or radiotherapy for this mantle cell lymphoma
2. Concurrent active malignancies, with the exception of in situ carcinoma of the cervix and basal cell carcinoma of the skin.
3. Grade 3 or 4 cardiac failure and/or ejection fraction < 50.
4. Psychological, familial, sociological or geographical conditions that do not permit treatment and/or medical follow-up required to comply with the study protocol.
5. Patients with a known history of human immunodeficiency virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS).
6. Presence of hepatitis or hepatitis B virus (HBV) infection.
7. Pregnant or breast-feeding women.
8. Central Nervous System (CNS) involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Izidore S. Lossos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alderuccio JP, Saul EE, Iyer SG, Reis IM, Alencar AJ, Rosenblatt JD, Lossos IS. R-MACLO-IVAM regimen followed by maintenance therapy induces durable remissions in untreated mantle cell lymphoma - Long term follow up results. Am J Hematol. 2021 Jun 1;96(6):680-689. doi: 10.1002/ajh.26163. Epub 2021 Apr 7. PMID 33735476

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R-MACLO/IVAM Group
Started | 25
Completed | 22
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) among study participants. PFS is defined as the time in years from start of treatment to the earliest one of the following events: relapse (in patients who achieve complete response), disease progression (in patients with partial response or stable disease), or death. PFS will be evaluated by treating physician from staging Computed Tomography (CT) or Positron Emission Tomography (PET) scans.
Time Frame: Up to 12 years
Population: Participants that completed Cycles 1 and 2 of R-MACLO/IVAM induction therapy.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 22
years | 8 [3.4 to 11]

2. Primary Outcome: Progression-Free Survival (PFS) Rate at 5 Years Using Kaplan-Meier Method
Description: Progression-Free Survival (PFS) rate at 5 years estimated by the Kaplan-Meier method will be reported as percentage probability of participants alive without relapse or disease progression at 5 years after starting study therapy. PFS is defined as the time from start of treatment to the earliest one of the following events: relapse (in patients who achieve complete response), disease progression (in patients with partial response or stable disease), or death. PFS will be evaluated by treating physician from staging Computed Tomography (CT) or Positron Emission Tomography (PET) scans.
Time Frame: 5 years
Population: Participants that completed Cycles 1 and 2 of R-MACLO/IVAM induction therapy.
Measure: Number (95% Confidence Interval); unit: percentage probability at 5 years
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 22
percentage probability at 5 years | 57.1 [31.3 to 76.3]

3. Secondary Outcome: Overall Survival (OS) Rate at 5 Years Using Kaplan-Meier Method
Description: Overall Survival (OS) rate at 5 years estimated by the Kaplan-Meier method will be reported as percentage probability of survival beyond 5 years. OS is defined as elapsed time from start date of treatment to date of death from any cause. Alive participants will be censored at last date known to be alive.
Time Frame: 5 years
Population: Participants that completed Cycles 1 and 2 of R-MACLO/IVAM induction therapy.
Measure: Number (95% Confidence Interval); unit: percentage probability at 5 years
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 22
percentage probability at 5 years | 79.7 [54.2 to 91.9]

4. Secondary Outcome: Rate of Response to Study Therapy
Description: The rate of response to study therapy will be reported as the number of participants achieving complete response (CR), complete response/unconfirmed (CRu) or partial response (PR) to protocol therapy according to criteria assignable to Non-Hodgkin's Lymphoma (NHL). Response assessment will be done by CT and Positron emission tomography (PET) scans, and bone marrow biopsy/aspirate, if clinically indicated.
Time Frame: Up to 8 years
Population: Participants that completed Cycles 1 and 2 of R-MACLO/IVAM induction therapy and evaluated for response.
Measure: Count of Participants; unit: Participants
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 22
Participants
  Complete Response (CR) | 20
  Complete Response unconfirmed (CRu) | 0
  Partial Response (PR) | 2

5. Secondary Outcome: Number of Participants Experiencing Treatment-Related Serious Adverse Events During R-MACLO/IVAM Induction Therapy
Description: The number of participants experiencing treatment-related serious adverse events (SAEs) during R-MACLO/IVAM induction therapy. AEs and SAEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0, as evaluated by treating physician.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 25
Participants | 2

6. Secondary Outcome: Number of Participants Experiencing Treatment-Related Adverse Events During R-MACLO/IVAM Induction Therapy
Description: The number of participants experiencing treatment-related adverse events (AEs) during R-MACLO/IVAM induction therapy. AEs and SAEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0, as evaluated by treating physician.
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | R-MACLO/IVAM Group
Number analyzed (Participants) | 25
Participants
  Grade 1 and 2 AEs | 25
  Grade 3 or higher AEs | 24

ADVERSE EVENTS:
Time Frame: 12 years
Arm/Group | R-MACLO/IVAM Group
All-Cause Mortality (participants affected / at risk) | 7/25
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-MACLO/IVAM Group (N=25)
Chemo induced myelodysplastic syndromes (MDS)/acute myeloid leukemia (AML) (Blood and lymphatic system disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infection, Lung (pneumonia) (Infections and infestations) | 2 (2)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (2)
Joint Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-MACLO/IVAM Group (N=25)
Abdominal distention (Gastrointestinal disorders) | 2 (2)
Abdominal pain (General disorders) | 6 (9)
Agitation (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 15 (51)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 10 (27)
Allergic reaction (Immune system disorders) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (15)
Anorexia (Gastrointestinal disorders) | 6 (7)
Anxiety (Nervous system disorders) | 6 (13)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (4)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 11 (35)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (9)
Autoimmune reaction (Immune system disorders) | 2 (4)
Back pain (General disorders) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1)
Blood - Other (Blood and lymphatic system disorders) | 6 (53)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (General disorders) | 7 (10)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (5)
Chest wall pain (General disorders) | 3 (4)
Confusion (Nervous system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 16 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 1 (2)
Creatinine increased (Metabolism and nutrition disorders) | 10 (45)
Cystitis (Renal and urinary disorders) | 1 (2)
Decubitus (Skin and subcutaneous tissue disorders) | 1 (2)
Depression (Nervous system disorders) | 4 (4)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 6 (13)
Diarrhea (Gastrointestinal disorders) | 17 (37)
Dizziness (Nervous system disorders) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (21)
Edema limbs (Blood and lymphatic system disorders) | 9 (25)
Encephalopathy (Nervous system disorders) | 1 (1)
Esophageal pain (General disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Eye pain (General disorders) | 1 (1)
Fatigue (General disorders) | 18 (61)
Febrile neutropenia (Infections and infestations) | 14 (31)
Fever (General disorders) | 15 (53)
Flatulence (Gastrointestinal disorders) | 3 (3)
Flushing (Skin and subcutaneous tissue disorders) | 2 (5)
Gastritis (Gastrointestinal disorders) | 5 (11)
Glomerular filtration rate decreased (Metabolism and nutrition disorders) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Headache (General disorders) | 16 (46)
Heartburn (Gastrointestinal disorders) | 5 (6)
Hemoglobin (Blood and lymphatic system disorders) | 24 (468)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 7 (40)
Hemorrhage nasal (Vascular disorders) | 4 (11)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (3)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Hot flashes (Endocrine disorders) | 1 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 11 (34)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 20 (149)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 6 (7)
Hypertension (Cardiac disorders) | 4 (26)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 24 (257)
Hypocalcemia (Metabolism and nutrition disorders) | 23 (202)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (13)
Hypokalemia (Metabolism and nutrition disorders) | 22 (107)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (38)
Hyponatremia (Metabolism and nutrition disorders) | 15 (45)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (20)
Hypotension (Cardiac disorders) | 6 (9)
Infection - Other (Specify) (Infections and infestations) | 3 (5) — Upper Respiratory Infection
Infection, Anal/perianal (Infections and infestations) | 1 (1)
Infection, Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection, Mucosa (Infections and infestations) | 1 (1)
Infection, Skin (cellulites) (Infections and infestations) | 2 (2)
Infection, Urinary tract NOS (Infections and infestations) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (4)
Insomnia (General disorders) | 5 (7)
Involuntary movement (Nervous system disorders) | 1 (3)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Leukocytes (Blood and lymphatic system disorders) | 25 (510)
Leukoencephalopathy (Nervous system disorders) | 1 (3)
Liver dysfunction (Hepatobiliary disorders) | 1 (1)
Lymphedema-related fibrosis (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 22 (330)
Mucositis (Gastrointestinal disorders) | 22 (56)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (79)
Neck pain (General disorders) | 1 (1)
Neuralgia (General disorders) | 2 (2)
Neurology - Other (Nervous system disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 25 (349)
Neuropathy: Sensory (Nervous system disorders) | 8 (14) — Peripheral sensory neuropathy
Oral pain (General disorders) | 1 (1)
Petechiae (Vascular disorders) | 8 (10)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngolaryngeal pain (General disorders) | 4 (4)
Phlebitis infective (Infections and infestations) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 24 (472)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (17)
Rash (Skin and subcutaneous tissue disorders) | 14 (35)
Rectal pain (General disorders) | 1 (2)
Rigors/chills (General disorders) | 15 (24)
Sepsis (Infections and infestations) | 6 (11)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (6)
Sweating (General disorders) | 4 (6)
Syncope (Nervous system disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Ureteric hemorrhage (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (12)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (43)
Weight loss (General disorders) | 4 (5)
Metabolic/Lab - Other (Nervous system disorders) | 9 (222)
Weight gain (General disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 6 (8)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Rhinitis (Immune system disorders) | 7 (12)
Retinal detachment (Eye disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (2)
Pulmonary - Other(specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Mild Upper respiratory infection
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Phlebitis (Infections and infestations) | 1 (1)
Neuropathy: Motor (Nervous system disorders) | 1 (12) — Peripheral motor neuropathy
Neuropathy: Cranial (Nervous system disorders) | 1 (2) — Olfactory nerve disorder
Palpitations (Cardiac disorders) | 1 (1)
Pain of skin (General disorders) | 1 (4)
Pain in extremity (General disorders) | 1 (1)
Otitis, middle ear (Ear and labyrinth disorders) | 1 (1)
Oral hemorrhage (General disorders) | 1 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 2 (2)
Gastrointestinal - Other (Specify) (Gastrointestinal disorders) | 1 (1) — Intermittent belching
Gastrointestinal - Other (Specify) (Gastrointestinal disorders) | 1 (1) — Gastroesophageal Reflux Disease (GERD)
Flashing vision (Eye disorders) | 2 (2)
Eye Infection (Infections and infestations) | 1 (1)
External ear pain (General disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Constitutional Symptoms - Other (General disorders) | 1 (1)
Cardiac arrhymthia (Cardiac disorders) | 1 (1)
Buttock pain (General disorders) | 1 (2)
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (2) — Basophilia
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (2) — Decreased red blood cells (RBC)
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Elevated absolute neutrophils
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Hypoglobulinemia
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Increased white blood cells (WBC)
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Leukocytosis
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Lymphocytosis
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (2) — Monocytosis
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) — Thrombocytopenia
Bladder hemorrhage (Renal and urinary disorders) | 1 (2)
Atrial tachycardia (Cardiac disorders) | 1 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Allergy - Other (Immune system disorders) | 1 (1)
Infection - Other (Specify) (Infections and infestations) | 1 (1) — Abdominal Infection
Infection - Other (Infections and infestations) | 1 (1)
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 3 (3) — Elevated/high Beta-2
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 2 (4) — Elevated/high BUN
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Decreased hematocrit (HCT)
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Decreased serum protein
Induration (Skin and subcutaneous tissue disorders) | 1 (1)
Infection, Upper airway NOS (Infections and infestations) | 1 (2)
Kidney pain (General disorders) | 1 (1)
Lymph node pain (General disorders) | 1 (1)
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Increased Absolute Neutrophils
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (4) — Increased lactate dehydrogenase (LDH)
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 2 (3) — Transaminitis
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Hypertriglyceridimia
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Hypocapnia
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 1 (1) — Hypochloremia
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 2 (4) — Hypercapnia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT00878254/Prot_SAP_000.pdf